CLINICAL TRIAL: NCT06132984
Title: Cardiac Magnetic Resonance Monitoring of Immune Checkpoint Inhibitor-related Cardiotoxicity in Patients With Gynecologic Malignancies: A Cohort Study
Brief Title: Cardiac Magnetic Resonance Monitoring of Immune Checkpoint Inhibitor-related Cardiotoxicity
Status: Recruiting | Type: Observational
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Ying-kun Guo, Professor, West China Second University Hospital
Other Study IDs: WestChinaSUH2022228
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Immune Checkpoint Inhibitors, Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with gynecologic malignancies who are preparing for ICIs treatment
  Interventions: Diagnostic Test: Cardiac magnetic resonance

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance — Cardiac magnetic resonance protocols include cine, non-contrast T1-mapping and T2-mapping.

SUMMARY:
This study is a prospective cohort clinical research that analyzes the changes in CMR parameters before and after immune checkpoint inhibitors (ICIs) therapy in patients with gynecologic malignancies. It also evaluates the value of CMR parameters in predicting long-term outcomes. The baseline assessment will be conducted prior to ICIs treatment, followed by multiple assessments during the medication process including within one week prior to cycle 3 , within the week prior to cycle 5 , 1 year after the first dose, and 2 years after the first dose. Assessment will also be conducted after discontinuation of ICIs medication. The assessment includes clinical assessment, CMR imaging, echocardiography, serum cardiac injury biomarkers, etc. Cancer therapy-related cardiac dysfunction (CTRCD), survival, and major adverse cardiac events (MACE) will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female patients aged 18 to 75 years, diagnosed with gynecological malignancies through histology or cytology.
* 2. Patients who are preparing for monotherapy or combination therapy with ICIs.
* 3. Voluntary signing of informed consent form.
* 4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* 5. Expected survival of at least 6 months.

Exclusion Criteria:

* 1. Previously received ICIs treatment.
* 2. With allergies or contraindications to ICIs.
* 3. Confirmed to be brain metastasis.
* 4. Patients who have major surgery within 4 weeks prior to or following the screening period.
* 5. Patients who have received systemic corticosteroids (at a dose equivalent to >10 mg prednisone per day) or other immunosuppressive medications within 14 days prior to enrollment or during the study period; however, the following situations are allowed for inclusion:

  1. the use of topical or inhaled corticosteroids is permitted;
  2. short-term (≤7 days) use of corticosteroids for prevention or treatment of non-autoimmune diseases is allowed.
* 6. Left ventricular ejection fraction (LVEF) ≤50%, or New York Heart Association functional classification (NYHA) ≥III.
* 7. Coronary heart disease, cardiomyopathy, congenital heart disease, valvular heart disease and pericardial diseases with confirmed diagnosis.
* 8. Lack of autonomous capacity, or a documented history of mental disease.
* 9. MRI contraindications: Pacemakers, neurostimulators, artificial metal heart valves, arterial aneurysm clips, intraocular metallic foreign bodies, inner ear implants, metal prostheses, metal limbs, metal joints, and any other metallic implants or foreign objects; severe hyperthermia patients; claustrophobia; severe respiratory conditions that prevent breath-holding.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with gynecologic malignancies who are preparing for ICIs treatment
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
cancer therapy-related cardiac dysfunction (CTRCD) | 2 month to 3 years
  Any reduction of LVEF to below 50% or a >10% reduction from baseline falling below the lower limit of normal.

SECONDARY OUTCOMES:
All-cause death; major adverse cardiac events (MACE) | 2 month to 3 years
  MACE were defined as a composite of cardiovascular death, cardiac arrest,cardiogenic shock, myocarditis, acute coronary syndromes (including non-ST-segment elevation and ST-segment elevation myocardial infarction), congestive heart failure, nonmalignant pericardial disorders, dysrhythmias（including complete heart block，documented sustained ventricular tachycardia, ventricular fibrillation)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang L, Zlotoff DA, Awadalla M, Mahmood SS, Nohria A, Hassan MZO, Thuny F, Zubiri L, Chen CL, Sullivan RJ, Alvi RM, Rokicki A, Murphy SP, Jones-O'Connor M, Heinzerling LM, Barac A, Forrestal BJ, Yang EH, Gupta D, Kirchberger MC, Shah SP, Rizvi MA, Sahni G, Mandawat A, Mahmoudi M, Ganatra S, Ederhy S, Zatarain-Nicolas E, Groarke JD, Tocchetti CG, Lyon AR, Thavendiranathan P, Cohen JV, Reynolds KL, Fradley MG, Neilan TG. Major Adverse Cardiovascular Events and the Timing and Dose of Corticosteroids in Immune Checkpoint Inhibitor-Associated Myocarditis. Circulation. 2020 Jun 16;141(24):2031-2034. doi: 10.1161/CIRCULATIONAHA.119.044703. Epub 2020 Jun 15. No abstract available. PMID 32539614
- [Background] Thavendiranathan P, Zhang L, Zafar A, Drobni ZD, Mahmood SS, Cabral M, Awadalla M, Nohria A, Zlotoff DA, Thuny F, Heinzerling LM, Barac A, Sullivan RJ, Chen CL, Gupta D, Kirchberger MC, Hartmann SE, Weinsaft JW, Gilman HK, Rizvi MA, Kovacina B, Michel C, Sahni G, Gonzalez-Mansilla A, Calles A, Fernandez-Aviles F, Mahmoudi M, Reynolds KL, Ganatra S, Gavira JJ, Gonzalez NS, Garcia de Yebenes Castro M, Kwong RY, Jerosch-Herold M, Coelho-Filho OR, Afilalo J, Zatarain-Nicolas E, Baksi AJ, Wintersperger BJ, Calvillo-Arguelles O, Ederhy S, Yang EH, Lyon AR, Fradley MG, Neilan TG. Myocardial T1 and T2 Mapping by Magnetic Resonance in Patients With Immune Checkpoint Inhibitor-Associated Myocarditis. J Am Coll Cardiol. 2021 Mar 30;77(12):1503-1516. doi: 10.1016/j.jacc.2021.01.050. PMID 33766256
- [Background] Cadour F, Cautela J, Rapacchi S, Varoquaux A, Habert P, Arnaud F, Jacquier A, Meilhac A, Paganelli F, Lalevee N, Scemama U, Thuny F. Cardiac MRI Features and Prognostic Value in Immune Checkpoint Inhibitor-induced Myocarditis. Radiology. 2022 Jun;303(3):512-521. doi: 10.1148/radiol.211765. Epub 2022 Mar 1. PMID 35230185
- [Background] Zhang L, Awadalla M, Mahmood SS, Nohria A, Hassan MZO, Thuny F, Zlotoff DA, Murphy SP, Stone JR, Golden DLA, Alvi RM, Rokicki A, Jones-O'Connor M, Cohen JV, Heinzerling LM, Mulligan C, Armanious M, Barac A, Forrestal BJ, Sullivan RJ, Kwong RY, Yang EH, Damrongwatanasuk R, Chen CL, Gupta D, Kirchberger MC, Moslehi JJ, Coelho-Filho OR, Ganatra S, Rizvi MA, Sahni G, Tocchetti CG, Mercurio V, Mahmoudi M, Lawrence DP, Reynolds KL, Weinsaft JW, Baksi AJ, Ederhy S, Groarke JD, Lyon AR, Fradley MG, Thavendiranathan P, Neilan TG. Cardiovascular magnetic resonance in immune checkpoint inhibitor-associated myocarditis. Eur Heart J. 2020 May 7;41(18):1733-1743. doi: 10.1093/eurheartj/ehaa051. PMID 32112560
- [Background] Faron A, Isaak A, Mesropyan N, Reinert M, Schwab K, Sirokay J, Sprinkart AM, Bauernfeind FG, Dabir D, Pieper CC, Heine A, Kuetting D, Attenberger U, Landsberg J, Luetkens JA. Cardiac MRI Depicts Immune Checkpoint Inhibitor-induced Myocarditis: A Prospective Study. Radiology. 2021 Dec;301(3):602-609. doi: 10.1148/radiol.2021210814. Epub 2021 Sep 28. PMID 34581628
- [Background] Liu J, Cao Y, Zhu K, Yao S, Yuan M, Kong X, Liu X, Li Y, Cui Y, Han X, Zhou X, Meng R, Shi H. Early evaluation of subclinical cardiotoxicity in patients with lung cancer receiving immune checkpoint inhibitors by cardiovascular magnetic resonance: a prospective observational study. Quant Imaging Med Surg. 2022 Oct;12(10):4771-4785. doi: 10.21037/qims-22-41. PMID 36185042
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455